CLINICAL TRIAL: NCT05782543
Title: Renal Ex Vivo Warm Advanced Resuscitation Through Machine Perfusion - The REWARM Study
Brief Title: Renal Ex Vivo Warm Advanced Resuscitation Through Machine Perfusion
Acronym: REWARM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15911
Record Dates: First submitted 2023-02-07; First posted 2023-03-23 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Kidney Transplant; Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypothermic machine perfusion (No Intervention)
- Normothermic machine perfusion (Active Comparator)
  Interventions: Procedure: Normothermic machine perfusion

INTERVENTIONS:
Procedure: Normothermic machine perfusion — To determine whether a 4-6 hour period of normothermic machine perfusion, following standard hypothermic machine perfusion, results in better graft function after transplantation, compared to hypothermic machine perfusion preservation alone of kidneys recovered from deceased donors aged 50 years or older
  Arms: Normothermic machine perfusion

SUMMARY:
The REWARM study is a randomized controlled clinical efficacy study, with primary outcome renal function 12 months after transplantation of kidneys recovered from deceased donors aged 50 years or older. Prior to transplantation, kidney grafts in the intervention group will receive 6 hours of NMP, following standard HMP and kidneys in the control group will only receive standard treatment, being HMP. It is a multi-center trial. Given the total annual 50+ deceased donor kidney transplantation volume of the three participating transplant centers combined, inclusions in the study are expected to last 2.5-3 years, aiming for a total of 120 patients in each of the two arms (240 patients total).

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving their first or second kidney transplant;
* Patients receiving a graft from a ≥ 50-year-old donor;
* Patients receiving a graft from a DCD or DBD donor;
* Patients receiving a kidney transplant in the UMCG, the Erasmus MC, or the LUMC;
* Patients receiving a graft stored on HMP;
* Patients ≥ 18 years of age;
* Patients having provided written informed consent.

Exclusion Criteria:

* Patients receiving their third or subsequent kidney transplant;
* Patients receiving a graft from a donor < 50 years;
* Patients receiving a graft not stored on HMP;
* Patients receiving a graft from a donor that underwent normothermic regional perfusion (NRP);
* Patients receiving a kidney transplant in another center than the UMCG, Erasmus MC, or LUMC;
* Patients receiving a multi-organ transplantation;
* Patients receiving a kidney with complex arterial anatomy (3 or more arteries);
* Recipients < 18 years of age.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Graft function at twelve months after transplantation | 12 months
  The primary endpoint of this study is graft function at twelve months after transplantation, defined as the estimated glomerular filtration rate (eGFR).

SECONDARY OUTCOMES:
Patient and graft survival | 12 months
  Patient and graft survival up to 12 months after transplantation
Occurence of delayed graft function (DGF) in the first 7 days after transplantation | 7 days
  DGF defined as dialysis requirement in the first week after transplantation, excluding dialysis for one-time hyperkaliemia in the first two days post-transplant
Duration of delayed graft function (DGF) in the first 7 days after transplantation | 7 days
  DGF defined as dialysis requirement in the first week after transplantation, excluding dialysis for one-time hyperkaliemia in the first two days post-transplant
Number of participants with primary non-function (PNF) | 12 months
  Incidence of primary non-function (PNF) defined as a permanent lack of graft function starting after transplantation.
Number of participants with biopsy-proven acute rejection | 12 monts
estimated Glomerular Filtration Rate | 12 months
  eGFR at day 7, and 1, 3, 6 and 12 months after transplantation
(serious) adverse events | 12 months
  Number of adverse (device) events and serious adverse (device) events
Postoperative complications | 12 months
The mean serum concentration of creatinine in umol/L for each study arm | 12 months
  Biochemical analysis of graft function with patient serum and urine levels of creatinine at postoperative day 0-7, and 1, 3, 6 and 12 months after transplantation
The mean serum concentration of urea in umol/L for each study arm | 12 months
  Biochemical analysis of graft function with patient serum and urine levels of urea at postoperative day 0-7, and 1, 3, 6 and 12 months after transplantation
The mean serum concentration of sodium in umol/L for each study arm | 12 months
  Biochemical analysis of graft function with patient serum and urine levels of sodium at postoperative day 0-7, and 1, 3, 6 and 12 months after transplantation
The mean serum concentration of potassium in umol/L for each study arm | 12 months
  Biochemical analysis of graft function with patient serum and urine levels of potassium at postoperative day 0-7, and 1, 3, 6 and 12 months after transplantation
The mean serum concentration of proteins in umol/L for each study arm | 12 months
  Biochemical analysis of graft function with patient serum and urine levels of protein at postoperative day 0-7, and 1, 3, 6 and 12 months after transplantation

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - University Medical Center Groningen, Groningen, Provincie Groningen
  - Leiden University Medical Center, Leiden
  - Erasmus Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Longchamp A, Markmann JF. Kidney Preservation Strategies to Improve Transplant Outcomes. Clin J Am Soc Nephrol. 2023 Dec 1;18(12):1628-1630. doi: 10.2215/CJN.0000000000000212. Epub 2023 May 23. No abstract available. PMID 37219010